CLINICAL TRIAL: NCT03827473
Title: ACADEMIC: A Randomized Phase II Clinical Trial of ADT Combined With Abiraterone or Docetaxel in Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Docetaxel or Abiraterone Acetate With ADT in Treating Patients With Metastatic Hormone Sensitive Prostate Cancer
Acronym: ACADEMIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was closed because the changing standard of care landscape, making this trial not impactful anymore.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI115099
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostatic Adenocarcinoma; Stage IV Prostate Cancer; Stage IVA Prostate Cancer; Stage IVB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Androgen Antagonists; Docetaxel; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (ADT, docetaxel) (Experimental): Participants receive androgen deprivation therapy (ADT) per standard of care and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antiandrogen Therapy; Drug: Docetaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (ADT, abiraterone acetate, prednisone) (Experimental): Participants receive androgen deprivation therapy (ADT) per standard of care, abiraterone acetate PO daily, and prednisone PO twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Antiandrogen Therapy; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
  Arms: Arm B (ADT, abiraterone acetate, prednisone)
Drug: Antiandrogen Therapy — Given per standard of care
  Other Names: ADT; Androgen Deprivation Therapy; Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm A (ADT, docetaxel)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
  Arms: Arm B (ADT, abiraterone acetate, prednisone)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well docetaxel or abiraterone acetate work when combined with androgen deprivation therapy (ADT) in treating patients with hormone sensitive prostate cancer that has spread to other parts of the body. Drugs used in chemotherapy, such as docetaxel and abiraterone acetate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Antihormone therapy, such as ADT may lessen the amount of androgen made by the body. It is not yet known whether docetaxel or abiraterone acetate work better when combined with ADT in treating patients with hormone sensitive prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of abiraterone acetate (abiraterone) and docetaxel on total quality of life between screening and month 12 of the study.

SECONDARY OBJECTIVES:

I. To assess prostate specific androgen (PSA) response rates across the entire population and compared between groups.

II. To assess impact of abiraterone and docetaxel on additional quality of life measurements and quality of life trends throughout the duration of the study.

III. To assess the potential clinical efficacy between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed adenocarcinoma of the prostate.
* Radiographically confirmed metastatic disease prior to patient enrollment. Metastatic disease can be confirmed based on conventional imaging (CT, MRI, nuclear medicine bone scan) or molecular imaging (fluciclovine-positron emission tomography (PET)/CT, prostate-specific membrane antigen (PSMA)-PET/CT, Choline-PET/CT etc).
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Absolute neutrophil count (ANC) >= 1.5 k/uL.
* Platelets >= 100 k/uL.
* Hemoglobin >= 9 g/dL.
* Serum total bilirubin =< 1.5 times upper limit of normal (ULN) OR direct bilirubin =< ULN for subjects with total bilirubin >= 1.5 x ULN.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 4 x ULN for subjects with liver metastases.
* Creatinine < 1.5 x ULN OR
* Creatinine clearance > 50 mL/min for subject with creatinine levels > 1.5 x ULN by Cockcroft-Gault formula or standard institutional practice.
* Highly effective method of contraception for both male and female partners of subjects throughout the study and for at least 3 months after last study treatment administration if the risk of conception exists.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically nonsignificant and/or stable on supportive therapy as defined by the treating physician.

Exclusion Criteria:

* No prior abiraterone or docetaxel therapy for metastatic hormone sensitive prostate cancer. Prior therapy with ADT or first generation anti-androgen receptor therapy (example: bicalutamide) is allowed.
* Completed any hormone therapy for localized prostate cancer and have recovery of testosterone (i.e. testosterone level is >50ng/dL).
* Patients have a histologic diagnosis of small cell prostate cancer or pure squamous cell prostate cancer.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias within 3 months of study enrollment.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 170 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack (TIA)), myocardial infarction (MI), or other ischemic event, or arterial thromboembolic event within 3 months before first dose.
  * Other clinically significant disorders that would preclude safe study participation. As defined by the treating physician.
* Known history of testing positive for human immunodeficiency virus (HIV) and cluster of differentiation 4 (CD4) count is below 200 or known acquired immunodeficiency syndrome diagnosis.
* Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or detectable HCV ribonucleic acid [RNA] if anti-HCV antibody screening test positive) and a detectable viral count at screening.
* Use of live virus vaccine within 4 weeks of the first dose of treatment or planned use while on trial for the duration of potential docetaxel treatment. Live vaccine use is acceptable after chemotherapy or for patients randomized to the abiraterone arm. There are no restrictions on inactive viruses.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (National Cancer Institute [NCI] CTCAE v5.0 grade >= 3).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maughan, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B (ADT, Abiraterone): Participants receive androgen deprivation therapy (ADT) per standard of care, abiraterone acetate PO daily, and prednisone PO twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Because only one participant enrolled, the baseline characteristics were not provided to protect the identify and privacy of the participant.
Groups:
- Arm A (ADT, Docetaxel): Participants receive ADT per standard of care and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
- Arm B (ADT, Abiraterone): Participants receive ADT per standard of care, abiraterone acetate PO daily, and prednisone PO twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life - FACT-P
Description: The impact of abiraterone acetate and docetaxel on health related quality of life will be assessed every 3 months from screening to month 12 of treatment or follow-up. The scale used will be the Functional Assessment of Cancer Therapy-Prostate (FACT-P) scale. The total score ranges from 0 to 156, with higher scores indicating a higher quality of life. The primary endpoint was intended to be quality of life at 12 months, but since no participants completed 12 months of treatment/follow-up, scores at baseline and 3 months are reported instead.
Time Frame: Planned for up to one year, but actual was 3 months
Population: There were no participants on Arm B to analyze.
Measure: Number; unit: score on a scale
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Number analyzed (Participants) | 1 | 0
score on a scale
  Baseline Score | 139.83 |
  Month 3 Score | 127 |

2. Secondary Outcome: Prostate-specific Antigen (PSA) Response
Description: PSA evaluations will occur every 3 months while on study. PSA response is defined as a reduction in PSA value of greater than or equal to 90% from baseline, reported as a count of participants who had a PSA response on the study.
Time Frame: Planned for up to 18 months, but actual was 3 months
Population: There were no participants on Arm B to analyze.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Number analyzed (Participants) | 1 | 0
Participants | 1 |

3. Secondary Outcome: Change in Quality of Life - FACT/GOG-NTX
Description: Quality of Life questionnaires will be done every 3 months while participants are on treatment. The scale used will be the Functional Assessment of Cancer Therapy (FACT)/Gynecologic Oncology Group (GOG)-Neurotoxicity (NTX) (FACT/GOG-NTX) scale (version 4). FACT/GOG-NTX total score ranges from 0 to 152, with higher scores indicating a higher quality of life.
Time Frame: Planned for up to 18 months, but actual was 3 months
Population: There were no participants on Arm B to analyze.
Measure: Number; unit: score on a scale
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Number analyzed (Participants) | 1 | 0
score on a scale
  Baseline Score | 131.83 |
  Month 3 Score | 126 |

4. Secondary Outcome: Change in Quality of Life - PROMIS Fatigue
Description: Quality of Life questionnaires will be done every 3 months while participants are on treatment. The scale used will be the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue scale. Total raw scores range from 7 to 35, with higher scores indicating a higher level of fatigue.
Time Frame: Planned for up to 18 months, but actual was 3 months
Population: There were no participants on Arm B to analyze.
Measure: Number; unit: score on a scale
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Number analyzed (Participants) | 1 | 0
score on a scale
  Baseline Score | 10 |
  Month 3 Score | 16 |

5. Secondary Outcome: Prostate Specific Antigen Progression Free Survival (PSA-PFS)
Description: Prostate Specific Antigen (PSA) will be measured every three months while on study. PSA Progression Free Survival (PSA-PSF) will be reported as the number of participants who have not demonstrated PSA progression by the end of the follow-up period. PSA progression is defined by meeting the following criteria: 1) an increase in PSA of greater than or equal to 25% from baseline or nadir, AND 2) an increase in PSA of at least 2 ng/dL, AND 3) the increase is confirmed at least 3 weeks later. This analysis was planned for up to 18 months following study enrollment, but the only participant enrolled on the study was only followed for 3 months.
Time Frame: Planned up to 18 months, but actual was 3 months
Population: There were no participants on Arm B to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
Number analyzed (Participants) | 1 | 0
Participants | 1 |

ADVERSE EVENTS:
Time Frame: Planned for up to 18 months, but due to low enrollment and early participant discontinuation, the actual time frame was 3 months.
Description: Information about adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, lab test or other means, were abstracted from clinic notes and recorded in the participant's study chart. The safety profile for the drugs involved in this study have been characterized extensively in previous clinical trials and standard clinical contexts. As such, safety data collection for this study was limited to ≥ Grade 3 adverse events.
Arm/Group | Arm A (ADT, Docetaxel) | Arm B (ADT, Abiraterone)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT03827473/Prot_SAP_000.pdf